CLINICAL TRIAL: NCT05281276
Title: A Phase Ib Study of Chidamide in Combination With Celecoxib in Patients With Metastatic Colorectal Cancer Who Had Progression or Were Intolerant of at Least Two Lines of Systemic Therapies (CCmCC)
Brief Title: Chidamide + Celecoxib in Advanced Metastatic Colorectal Cancer (CCmCC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The overall profile does not support development for metastatic colorectal cancer
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Chao Tsu-Yi, Director, Cancer Center, Taipei Medical University Shuang Ho Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: N202007026
Record Dates: First submitted 2021-11-15; First posted 2022-03-16 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; HBI-8000; Celecoxib

STUDY DESIGN:
Intervention Model Description: Cohort1: Chidamide(20mg)+Celecoxib(200mg); Cohort2: Chidamide(30mg)+Celecoxib(200mg)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chidamide (20 mg) BIW in combination with celecoxib (CC) (Experimental): Chidamide: The dosing schedule is four/six tablets (20 mg) BIW, taken at 30 min after breakfast. The interval between two doses in each week should not be less than 3 days.
  Celecoxib: The dosing schedule is one capsule (200 mg) daily taken at 30 min after breakfast.
  A treatment cycle is defined as a period of 4 weeks (28 days)
  Interventions: Drug: chidamide; Drug: celecoxib
- chidamide(30 mg) BIW in combination with celecoxib (CC) (Experimental): Chidamide: The dosing schedule is four/six tablets (30 mg) BIW, taken at 30 min after breakfast. The interval between two doses in each week should not be less than 3 days.
  Celecoxib: The dosing schedule is one capsule (200 mg) daily taken at 30 min after breakfast.
  A treatment cycle is defined as a period of 4 weeks (28 days)
  Interventions: Drug: chidamide; Drug: celecoxib

INTERVENTIONS:
Drug: chidamide — During the run-in period, the patients will take a single dose of chidamide on Day 3. In a 28-day treatment cycle, the dosing schedule is four/six table (20/30mg) BIW .
  Other Names: tucidinostat; HBI-8000
Drug: celecoxib — During the run-in period, the patients will take a single dose of celecoxib on Day 1. In a treatment cycle, the dosing schedule is one capsule(200 mg) daily.
  Other Names: Celebrex

SUMMARY:
This study is designed as an open-label, dose-escalation manner to determine the MFD of chidamide in combination with celecoxib in patients with advanced mCRC.

DETAILED DESCRIPTION:
This is a monocentric, open-label, non-randomized dose feasibility study trial to characterize the safety, tolerability, pharmacokinetics, and preliminary efficacy of chidamide in combination with celecoxib in patients with advanced mCRC. Each cohort will have up to 6 subjects. Eligible patients will be assigned to 1 of up to 2 sequential cohorts. The planned dose levels of the two cohorts include (1) 20 mg chidamide plus 200 mg celecoxib; and (2) 30 mg chidamide plus 200 mg celecoxib.

For each subject, the treatment period is divided into two periods, a run-in period and a combination therapy period.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is 20-year-old or older on the day that consent is provided.
2. With histologically or cytologically proven metastatic colorectal adenocarcinoma.
3. Have measurable lesions according to RECIST v1.1.
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 to 2.
5. Adequate organ function as defined below:

   i. White blood cells (WBC) ≥3,000/μL ii. Absolute neutrophil count ≥1,500/μL iii. Platelets ≥1 x 105/μL iv. Hemoglobin ≥9.0 g/dL v. Total bilirubin ≤1.5 x the upper limit of normal (ULN) vi. AST(SGOT)/ALT(SGPT) ≤3 x ULN (or ≤5 x ULN if liver metastases are present) vii. Serum creatinine ≤1.5 x ULN
6. Patients who had received or were intolerant of at least 2 front-line systemic treatments. In addition, patients have failed or refused all available standard treatment, or were intolerant of such treatments. For K-ras wild type tumor, anti-EGFR therapy must have been done. For K-ras mutant tumor, antiangiogenic therapy must have been done.
7. Able to take oral medication.
8. With a life expectancy of at least 3 months.
9. Female patients of childbearing potential must have a negative urine or serum pregnancy test.
10. Patients in reproductive age must be willing to use adequate contraception (refer to Section 8.4.2 of the protocol for adequate contraception methods) during the study and 3 months after the end of the study.
11. Ability to understand and the willingness to provide a written informed consent document.

Exclusion Criteria:

(I) Inclusion criteria:

1. The patient is 20-year-old or older on the day that consent is provided.
2. With histologically or cytologically proven metastatic colorectal adenocarcinoma.
3. Have measurable lesions according to RECIST v1.1.
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 to 2.
5. Adequate organ function as defined below:

   i. White blood cells (WBC) ≥3,000/μL ii. Absolute neutrophil count ≥1,500/μL iii. Platelets ≥1 x 105/μL iv. Hemoglobin ≥9.0 g/dL v. Total bilirubin ≤1.5 x the upper limit of normal (ULN) vi. AST(SGOT)/ALT(SGPT) ≤3 x ULN (or ≤5 x ULN if liver metastases are present) vii. Serum creatinine ≤1.5 x ULN
6. Patients who had received or were intolerant of at least 2 front-line systemic treatments. In addition, patients have failed or refused all available standard treatment, or were intolerant of such treatments. For K-ras wild type tumor, anti-EGFR therapy must have been done. For K-ras mutant tumor, antiangiogenic therapy must have been done.
7. Able to take oral medication.
8. With a life expectancy of at least 3 months.
9. Female patients of childbearing potential must have a negative urine or serum pregnancy test.
10. Patients in reproductive age must be willing to use adequate contraception (refer to Section 8.4.2 of the protocol for adequate contraception methods) during the study and 3 months after the end of the study.
11. Ability to understand and the willingness to provide a written informed consent document.

(II) Exclusion criteria:

1. With known central nervous system (CNS) metastases, a history of CNS metastases or leptomeningeal diseases.
2. With known hypersensitivity towards chidamide, celecoxib, sulfonamides, aspirin, NSAIDs, or any other agents used in the study, including the excipient in the study agent; or with history of asthma, urticarial, or other allergic-type reactions after taking aspirin or other NSAIDs.
3. With severe systemic disease, such as renal disease (serum creatinine >1.5 x ULN), liver disease (AST/ALT >3 x ULN, AST/ALT >5 x ULN if metastatic liver disease were known), active gastrointestinal hemorrhage or increased risks of gastrointestinal bleeding, uncontrolled diabetes, or uncontrolled hypertension.
4. With uncontrolled or significant cardiovascular diseases, including:

   i. Symptomatic congestive heart failure within 6 months prior to screening, or left ventricular ejection fraction <50% prior to screening ii. Myocardial infarction within 12 months prior to screening iii. Severe or unstable angina within 6 months prior to screening iv. History of any significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, or TdP) v. History of significant QT interval prolongation, or corrected QT interval (QTc) >450 ms prior to screening vi. History of cerebrovascular accident vii. Symptomatic coronary heart disease requiring treatment with agents
5. With the size of fluid area detected by cardiac ultrasonography in cavum pericardium ≥ 10 mm.
6. With history of organ transplantation.
7. With known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
8. With autoimmune disorders or history of organ transplantation who require immunosuppressive therapy.
9. Has had prior chemotherapy, targeted small molecule therapy, radiation therapy, or any NSAID within 2 weeks prior to the first dose of study medication or who has not recovered from adverse events to CTCAE v5.0 Grade 1 due to a previously administered agent.
10. Has clinical significant gastrointestinal abnormality, e.g., unable to swallow, chronic diarrhea, ileus, or bowel obstruction, which would interfere the ingestion, transportation, or absorption of oral agents.
11. With active infection [suffered from active infection of bacteria, virus, fungi, mycobacteria, parasites, or other infections (excluding nail bed fungal infections), or require intravenous antibiotic therapy, or antiviral therapy, or hospitalization due to any significant infection events within 4 weeks], or persistent fever within 14 days prior to study entry.
12. Had major surgery <6 weeks prior to study entry.
13. Has known psychiatric disorder, mental deficiency, or substance abuse disorder that would limit compliance with study requirements.
14. Is currently participating and receiving study therapy, or has participated in a study of an investigational agent and received study therapy or used an investigation device within 4 weeks of the first dose of study medication.
15. Pregnant or lactating female.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might interfere the results of the trial or is not in the best interest of the subject to participate, in the opinion of the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Maximum Feasible Dose (MFD) | defined as the highest dose for which ≤1 of 6 evaluable subjects experiencing DLT during the first treatment cycle (28 days) of the combination therapy, assessed up to 24 months
  Maximum Feasible Dose (MFD): is defined as the highest dose for which ≤1 of 6 evaluable subjects experiencing DLT during the first treatment cycle (28 days) of the combination therapy. If the dose of Cohort 1 is not tolerable by ≥2 evaluable subjects, the MFD will be considered as not determined.
Pharmacokinetics profiles-(AUC0-t) | Run-in period, on day1, blood sample will be 0, 1, 2, 6, 12, and 24 hours; on day3, blood sample will be 0, 1, 2, 6, 12, 24, 48, and 72 hours.Combination therapy period, on day1 & day25, blood sample will be 0, 1, 2, 6, 12, 24, 48 and 72 hours.
  Area under the plasma concentration-time curve from time zero to time t(AUC0-t)
Pharmacokinetics profiles-(AUC0-∞) | Run-in period, on day1, blood sample will be 0, 1, 2, 6, 12, and 24 hours; on day3, blood sample will be 0, 1, 2, 6, 12, 24, 48, and 72 hours.Combination therapy period, on day1 & day25, blood sample will be 0, 1, 2, 6, 12, 24, 48 and 72 hours.
  Area under the plasma concentration-time curve from time zero to infinity(AUC0-∞)
Pharmacokinetics profiles-(Cmax) | Run-in period, on day1, blood sample will be 0, 1, 2, 6, 12, and 24 hours; on day3, blood sample will be 0, 1, 2, 6, 12, 24, 48, and 72 hours.Combination therapy period, on day1 & day25, blood sample will be 0, 1, 2, 6, 12, 24, 48 and 72 hours.
  Maximum plasma concentration(Cmax)
Pharmacokinetics profiles-(Tmax) | Run-in period, on day1, blood sample will be 0, 1, 2, 6, 12, and 24 hours; on day3, blood sample will be 0, 1, 2, 6, 12, 24, 48, and 72 hours.Combination therapy period, on day1 & day25, blood sample will be 0, 1, 2, 6, 12, 24, 48 and 72 hours.
  Time to maximum plasma concentration(Tmax)
Pharmacokinetics profiles-(T1/2) | Run-in period, on day1, blood sample will be 0, 1, 2, 6, 12, and 24 hours; on day3, blood sample will be 0, 1, 2, 6, 12, 24, 48, and 72 hours.Combination therapy period, on day1 & day25, blood sample will be 0, 1, 2, 6, 12, 24, 48 and 72 hours.
  Half-life(T1/2)
Pharmacokinetics profiles-(Kel) | Run-in period, on day1, blood sample will be 0, 1, 2, 6, 12, and 24 hours; on day3, blood sample will be 0, 1, 2, 6, 12, 24, 48, and 72 hours.Combination therapy period, on day1 & day25, blood sample will be 0, 1, 2, 6, 12, 24, 48 and 72 hours.
  Elimination rate constant(Kel)
Pharmacokinetics profiles-(AUC0-τ,ss) | Run-in period, on day1, blood sample will be 0, 1, 2, 6, 12, and 24 hours; on day3, blood sample will be 0, 1, 2, 6, 12, 24, 48, and 72 hours.Combination therapy period, on day1 & day25, blood sample will be 0, 1, 2, 6, 12, 24, 48 and 72 hours.
  Area under the plasma concentration-time curve from time zero to time τ (dosing interval) at steady state(AUC0-τ,ss)
Pharmacokinetics profiles-(Cave,ss) | Run-in period, on day1, blood sample will be 0, 1, 2, 6, 12, and 24 hours; on day3, blood sample will be 0, 1, 2, 6, 12, 24, 48, and 72 hours.Combination therapy period, on day1 & day25, blood sample will be 0, 1, 2, 6, 12, 24, 48 and 72 hours.
  Average plasma concentration at steady state(Cave,ss)
Pharmacokinetics profiles-(Cmin,ss) | Run-in period, on day1, blood sample will be 0, 1, 2, 6, 12, and 24 hours; on day3, blood sample will be 0, 1, 2, 6, 12, 24, 48, and 72 hours.Combination therapy period, on day1 & day25, blood sample will be 0, 1, 2, 6, 12, 24, 48 and 72 hours.
  Minimum (trough) plasma concentration at steady state(Cmin,ss)
Pharmacokinetics profiles-(Cmax,ss) | Run-in period, on day1, blood sample will be 0, 1, 2, 6, 12, and 24 hours; on day3, blood sample will be 0, 1, 2, 6, 12, 24, 48, and 72 hours.Combination therapy period, on day1 & day25, blood sample will be 0, 1, 2, 6, 12, 24, 48 and 72 hours.
  Maximum (peak) plasma concentration at steady state(Cmax,ss)
Pharmacokinetics profiles-(Tmax,ss) | Run-in period, on day1, blood sample will be 0, 1, 2, 6, 12, and 24 hours; on day3, blood sample will be 0, 1, 2, 6, 12, 24, 48, and 72 hours.Combination therapy period, on day1 & day25, blood sample will be 0, 1, 2, 6, 12, 24, 48 and 72 hours.
  Time to maximum plasma concentration at steady state(Tmax,ss)
Pharmacokinetics profiles-(DF) | Run-in period, on day1, blood sample will be 0, 1, 2, 6, 12, and 24 hours; on day3, blood sample will be 0, 1, 2, 6, 12, 24, 48, and 72 hours.Combination therapy period, on day1 & day25, blood sample will be 0, 1, 2, 6, 12, 24, 48 and 72 hours.
  Degree of fluctuation(DF)

SECONDARY OUTCOMES:
Progression-free survival | from the time of first day of dosing (Run-in period Day1) until the date of first objective disease progression or death, assessed up to 24 months
  defined as the time from first day of dosing until the date of first objective disease progression or death. Patients who have not progressed or died at the time of analysis will be censored at the time of the latest date of tumor assessment
Objective response | From enrollment until disease progression or unacceptable toxicity, assessed up to 24 months
  ORR, defined as the percentage of patients with CR and PR of total number of analysis set

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Undecided